CLINICAL TRIAL: NCT06046469
Title: Validity of Computed Tomography Versus Magnetic Resonance Imaging in Predicting Muscular Invasion of Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abdulrhman Ismail Abdulrhman Elkhouly, Abdulrahman Ismail Elkhouly, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CT vs MRI in bladder cancer
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT group (Active Comparator): this group of patient is doing CT abdomen and plevis with IV contrast then they undergo TURBT and compare the radiological staging to histopathological staging.
  Interventions: Diagnostic Test: CT with contrast; Procedure: TURBT
- MRI group (Active Comparator): this group of patient is doing MRI pelvis with contrast then they undergo TURBT and compare the radiological staging to histopathological staging.
  Interventions: Diagnostic Test: MRI pelvis; Procedure: TURBT

INTERVENTIONS:
Diagnostic Test: CT with contrast — CT abdomen and pelvis with IV contrast
  Arms: CT group
Diagnostic Test: MRI pelvis — MRI pelvis with contrast
  Arms: MRI group
Procedure: TURBT — transurethral resection of bladder tumor

SUMMARY:
The aim of this work is to compare validity between CT and MRI in detecting muscular invasion in Patients with bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with urinary bladder mass

Exclusion Criteria:

* bleeding tendency ,patients had chemo , radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
which is better to detect muscular invasion in bladder cancer CT vs MRI | 1 month
  the radiological staging of CT and MRI compared to histopathological staging

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Menofia University, Shibīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No